CLINICAL TRIAL: NCT04824144
Title: Effects of Dexmedetomidine in Patients With Agitated Delirium in Palliative Care: an Open-label Phase 1/2 Proof-of-concept, Feasibility, and Dose-finding Clinical Trial
Brief Title: Effects of Dexmedetomidine in Patients With Agitated Delirium in Palliative Care
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bruyère Health Research Institute. (Other)
Collaborators: The Ottawa Hospital (Other); Bruyère Continuing Care (Unknown); Foothills Medical Centre (Other)
Responsible Party: Principal Investigator, James Downar, Head, Division of Palliative Care, Bruyère Health Research Institute.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 339633386643463
Record Dates: First submitted 2021-03-22; First posted 2021-04-01 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-08

CONDITIONS: Hyperactive Delirium; Delirium of Mixed Origin
Keywords: Dexmedetomidine; Agitation; Delirium; Palliative; End of life
MeSH Terms: conditions — Delirium; Psychomotor Agitation; Death | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: The study is a multi-site, open-label, single-arm phase 1/2 proof-of-concept, dose-finding, feasibility, and preliminary efficacy clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dexmedetomidine subcutaneous continuous infusion (Experimental): Participants will be given a starting low dose of 0.4 mcg/kg/hr, to be titrated up to a medium dose of 0.7 mcg/kg/hr and potentially up to a maximum dose of 1.0 mcg/kg/hr by subcutaneous infusion until the target RASS-PAL level has been achieved.
  Interventions: Drug: Dexmedetomidine Hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Dexmedetomidine will be administered by subcutaneous continuous infusion using a Continuous Ambulatory Delivery Device (CADD pump).
  Other Names: Dexmedetomidine; Precedex

SUMMARY:
The goal of this multi-centre phase I/II open-label, single-arm study is to determine the feasibility, optimal dose, and preliminary efficacy of dexmedetomidine to manage agitated delirium among patients near the end of life followed by a palliative care provider in a non-monitored setting. Fifty patients will receive dexmedetomidine (0.4 mcg/kg/hour, titrated up to 1.0 mcg/kg/hour) subcutaneously. Feasibility (recruitment rate, cost), safety (rate of adverse events), dosing, and preliminary efficacy (agitation, delirium severity) will be measured.

DETAILED DESCRIPTION:
Delirium is a common and challenging complication to manage at the end of life. An estimated 75% (range 58-88%) of patients experience delirium during a palliative inpatient admission in the weeks prior to death. Delirium is classified on the basis of psychomotor activity into hypoactive, hyperactive, and mixed subtypes. Agitation is a feature of both the hyperactive and mixed subtypes and, when present, the episode of delirium is conventionally referred to as agitated delirium. Agitated delirium is characterized by increased agitation, verbal or physical aggression, and perceptual disturbance. Furthermore, these episodes can cause the patient, their families, and the care team significant distress by decreasing a patient's ability to communicate with loved ones and the care team. Studies of patients who recall their delirium experience during an inpatient hospital admission report high levels of distress, and that this distress is exacerbated by being aware of their inability to communicate with family and the healthcare team.

However, studies demonstrate distress associated with delirium is greater among family members compared to that experienced by patients. In the context of palliative care, agitated delirium in the dying phase is particularly devastating for family members - the inability to meaningfully communicate with a loved one during final interactions with them, and to witness the visible distress that characterizes agitated delirium, can cause significant anguish. Several studies demonstrate severe levels of distress among a majority of caregivers who have cared for a loved one with delirium. Family members of patients with terminal delirium report negative physical and psychological burden associated with delirium, including family member feelings of distress, anxiety, and helplessness, exhaustion, and difficulty coping. Additionally, caregiver-perceived delirium in the last 6 months of life has been found to be associated with significantly increased risk - up to 12x - of symptoms of generalized anxiety among family caregivers. In particular, patient symptoms characteristic of agitated delirium, such as restlessness and agitation, psychotic symptoms, cognitive impairment, and communication difficulties, are associated with greater levels of psychological and emotional distress among family members. Bereaved family members express experiencing anger and sadness that they could not have meaningful interactions with their loved one at the end of life, and felt delirium robbed them prematurely of these interactions before death and hindered their opportunity to say goodbye. Family members have further described this phenomenon as distress related to premature loss of the caregiver-patient relationship and the loss of a familiar person becoming a stranger. Family members also report distress related to decision-making that balances their desire for meaningful communication at the end of life with reducing patient suffering. Most commonly, this dilemma is manifested in family member decisions around the use of sedation.

Agitated delirium also has a marked impact on nursing staff and their ability to assess patient needs. Qualitative investigations of palliative care nurses' experiences caring for patients with delirium found nurses had difficulty managing patient delirium in a way they felt maintained patients' dignity and "minimized chaos", and reported delirium and related symptoms were highly distressing for them. Specifically, delirium-related distress experienced by nurses has been shown to be significantly associated with patient delirium severity and the presence and severity of perceptual disturbances. Clinical professionals have also expressed negative effects of delirium on their interactions with family members, with disagreements and tension arising from different understandings of patient needs.

There is limited evidence to support the use of pharmacological interventions for the management of delirium symptoms in palliative care patients, and no medication currently approved in Canada for the indication of delirium. However, published guidelines do recognize a limited role for the use of medications (such as low doses of antipsychotics and/or benzodiazepines) in distressed delirious patients or if there are safety concerns. Among imminently dying patients, pharmacological sedation (e.g., with midazolam, methotrimeprazine, or phenobarbital) is often used to manage agitated delirium; however, use of these medications to manage delirium in the dying phase is based on case series and expert opinion. More broadly, clinical guidelines and systematic reviews of palliative pharmacological sedation conclude that evidence for the efficacy of sedation for symptom control using these medications is insufficient. Additionally, sedation to treat agitated delirium is limited in that it generally eliminates patients' ability to be alert and interact with others, a limitation that, as outlined above, is often contrary to patients' goals of care and the well-being of family members. There is a need for alternative interventions that better align with patients' goals of care and support patients, family members, and clinical staff through meaningful communication at the end of life.

An increasing number of small case series and reviews suggest dexmedetomidine may be an effective and safe option for managing agitated delirium in palliative care. Dexmedetomidine is a centrally active alpha-2 receptor agonist that has mild sedative and opioid co-analgesic effects without suppressing respiratory drive. In most acute care hospital settings, dexmedetomidine is restricted for use in the intensive care unit and by anesthesia for short term sedation. Delirium treatment and prevention has commonly been studied as a secondary endpoint in clinical trials of sedation for critically ill patients, largely demonstrating the effectiveness of dexmedetomidine for delirium management over currently used medications in palliative care, including haloperidol, midazolam, and propofol. Given dexmedetomidine is currently the only agent recommended for treatment of agitated delirium in critically ill patients, pilot data reports have emerged regarding its use in other settings where agitated delirium is highly prevalent, namely palliative care. The largest and most recent case series (n=6) of dexmedetomidine to manage agitated delirium reported improved patient agitation and distress in all cases while maintaining a rousable, conscious state, providing patients the opportunity to interact with others at the end of life. Similarly, additional case studies of agitated delirium in palliative care (total n=4) have all reported successful resolution and/or symptom control of patients' agitated delirium at the end of life. In terms of dosage, these therapeutic benefits were predominantly achieved with moderate to high doses of dexmedetomidine (e.g., 0.5 mcg/kg/hr-1.5 mcg/kg/hr). Similarly, initial findings from our unpublished retrospective case series of dexmedetomidine to manage agitated delirium in palliative care (n=10) revealed moderate success at dose levels of 0.4 mcg/kg/hr-0.7 mcg/kg/hr, but minimal success at low dose levels of 0.2 mcg/kg/hr-0.3 mcg/kg/hr.

In contrast to other medications commonly used to manage agitated delirium, dexmedetomidine provides rousable sedation, better supporting communication needs and goals of care at the end of life. Dexmedetomidine is now off-patent, reducing previous cost barriers to use. In addition, while dexmedetomidine is administered intravenously in critical care, advance preparation for subcutaneous administration is more conducive to use in palliative care. To facilitate this, our team recently completed stability testing and demonstrated >90% retention of dexmedetomidine 20mcg/ml in 0.9% sodium chloride in polyvinylchloride bags after 9 days of storage at both room temperature (25°C ± 2°C) and refrigeration (4°C ± 2°C ) (accepted for publication). Furthermore, evidence demonstrates subcutaneous administration of dexmedetomidine results in a relative bioavailability of about 80%.

The investigators propose to evaluate the safety, feasibility, and preliminary efficacy of dexmedetomidine for the management of agitated delirium in palliative care. There are currently no approved therapies for agitated delirium in palliative care, but evidence from critical care, reduced medication costs, and published case series in palliative care suggest dexmedetomidine may be effective to treat this challenging condition. A therapy that might treat delirium without causing excess sedation, allowing patients to continue interactions with their loved ones and care team, would be a "game changer" in palliative care. There is the potential to improve end-of-life care for patients and their families in a manner that is more consistent with their goals of care and provides necessary symptom management while reducing the distress experienced by family and healthcare team members.

Details of Eligibility, Intervention Protocol, and Outcome Measures are provided elsewhere.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years)
2. Admitted to a participating inpatient palliative care unit
3. Meeting one of the following criteria:

   1. Agitated delirium: (i) Richmond Agitation-Sedation Scale for palliative care patients (RASS-PAL) score of +2 or greater and (ii) Confusion Assessment Method (CAM) positive status and (iii) Without a known potentially reversible cause (e.g. hypercalcemia, specific medication infection, etc.), or in whom the patient/Substitute Decision Maker (SDM) has requested not to treat the cause.
   2. Previous history of delirium (in the last 6 months)
   3. Patient is within the last two weeks of life and is expected to die during this admission (MRP judgement)

Exclusion Criteria:

1. Hemodynamic instability (systolic blood pressure <80mmHg)
2. Bradyarrhythmia (heart rate < 60) at baseline
3. Patients on verapamil, diltiazem, or beta-blocker (patients are eligible if these medications are stopped prior to receiving dexmedetomidine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Dosing - Therapeutic Dose | Enrollment to study withdrawal, hospital discharge, or death, whichever is first
  Dose at which the target Richmond Agitation Sedation Scale-Palliative (RASS-PAL) score of -1 ("drowsy"), 0 ("alert and calm"), or +1 ("restless") is achieved. The RASS-PAL is a 10-point scale with scores ranging from -5 (not rousable) to +4 (combative).
Dosing - Time | Enrollment to study withdrawal, hospital discharge, or death, whichever is first
  Time (in hours) at which the target Richmond Agitation Sedation Scale-Palliative (RASS-PAL) score of -1 ("drowsy"), 0 ("alert and calm"), or +1 ("restless") is achieved. The RASS-PAL is a 10-point scale with scores ranging from -5 (not rousable) to +4 (combative).
Number of Participants With Adverse Events - Bradycardia | Enrollment to study withdrawal, hospital discharge, or death, whichever is first
  Proportion of participants with Bradycardia (two consecutive readings of heart rate (HR)<40 beats/minute)
Number of Participants With Adverse Events - Hypotension | Enrollment to study withdrawal, hospital discharge, or death, whichever is first
  Proportion of participants with Hypotension (systolic blood pressure(SBP) < 70 mmHg or 40% drop from baseline with lightheadedness or loss of consciousness.
Number of Participants With Adverse Events - Skin Tolerability | Enrollment to study withdrawal, hospital discharge, or death, whichever is first
  Proportion of participants with skin intolerability of the infusion site, based on the National Cancer Institute Common Toxicity for Adverse Events.
Recruitment Rate | Through study completion, up to 1 year
  Number of patients enrolled divided by number of patients approached.
Cost | Through study completion, up to 13 months
  Comparison of total drug cost of dexmedetomidine (accounting for total dosage administered and duration of therapy) and compare the total cost to that of the alternative first line sedative identified by the treating physician.
Baseline Agitation | Baseline
  Measured using the Richmond Agitation Sedation Scale-Palliative (RASS-PAL). The RASS-PAL is a 10-point scale with scores ranging from -5 (not rousable) to +4 (combative).
Baseline Delirium Severity | Baseline
  Measured using the Nursing Delirium Screening Tool (Nu-DESC). Nu-DESC scores range from 0 to 10, with higher scores indicating worse delirium.
Change in Agitation | Measured at Day 1 - 1 hour post administration, one hour post any dose change, and once daily from Day 1 to intervention completion (up to 13 months)
  Measured using the Richmond Agitation Sedation Scale-Palliative (RASS-PAL). RASS-PAL is a 10-point scale with scores ranging from -5 (not rousable) to +4 (combative).
Change in Delirium Severity | Measured every 8 hours from Day 1 to intervention completion (up to 13 months)
  Measured using the Nursing Delirium Screening Tool (Nu-DESC). Nu-DESC scores range from 0 to 10, with higher scores indicating worse delirium.

SECONDARY OUTCOMES:
Baseline Pain | Baseline
  Measured using the Critical Care Pain Observation Tool (CPOT) (higher score indicates worse pain).
Change in Pain From Baseline | Measured once daily from Day 1 to intervention completion (up to 13 months)
  Measured using the Critical Care Pain Observation Tool (CPOT) (higher score indicates worse pain).
Baseline Opioid Use | Measured at Baseline
  Measured using the oral Morphine-Equivalent Daily Dose (MEDD) and frequency of breakthrough dose for each participant
Change in Opioid Use From Baseline | Measured once daily from Day 1 to intervention completion (up to 13 months)
  Measured using the oral Morphine-Equivalent Daily Dose (MEDD) and frequency of breakthrough dose for each participant

CONTACTS AND LOCATIONS:
Overall Officials: James Downar, MDCM, MSc, Principal Investigator — Bruyère Health Research Institute.
Locations (3):
- Canada (3):
  - Foothills Medical Centre, Calgary, Alberta
  - The Ottawa Hospital, Ottawa, Ontario
  - Bruyère Continuing Care, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No